CLINICAL TRIAL: NCT05278104
Title: Double-blind, Randomized, Parallel Group, Placebo Controlled Clinical Trial to Evaluate the Effects of Atomoxetine on Impulsivity in Behavioral Laboratory Tasks in Adult ADHD Patients
Brief Title: A Study to Test Different Ways to Measure the Effect of Atomoxetine on Impulsive Behavior in Young Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0352-2159; 2021-005270-26 (EudraCT Number)
Record Dates: First submitted 2022-03-11; First posted 2022-03-14 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atomoxetine (Experimental): Day 1 and Day 8:
  After fasting for at least 10 hours overnight, participants received a single dose of Atomoxetine consisting of two 40 mg capsules (totaling 80 mg) in the morning at the trial site.
  Day 2 to Day 7:
  Participants took a single dose of Atomoxetine consisting of one 40 mg capsule in the morning at home.
  Day 9 to Day 14:
  Participants took a single dose of Atomoxetine consisting of two 40 mg capsules (totaling 80 mg) in the morning at home.
  Interventions: Drug: Zentiva®
- Placebo (matching Atomoxetine) (Placebo Comparator): Day 1 and Day 8:
  After fasting for at least 10 hours overnight, participants received a single dose of placebo (matching Atomoxetine) in the morning at the trial site.
  Day 2 to Day 7:
  Participants took a single dose of placebo (matching Atomoxetine) in the morning at home.
  Day 9 to Day 14:
  Participants took a single dose of placebo (matching Atomoxetine) in the morning at home.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zentiva® — Zentiva®, oral, tablet
  Other Names: Atomoxetin
  Arms: Atomoxetine
Drug: Placebo — Placebo, oral, tablet
  Arms: Placebo (matching Atomoxetine)

SUMMARY:
The primary objectives are to investigate the effect of atomoxetine on impulsivity after single dose and at steady state measured by the total score of Barrett Impulsiveness Scale version 11 (BIS-11) and Short Urgency, Perseverance, Premeditation, and Sensation Seeking-Positive Urgency Impulsive Behavior Scale (S-UPPS-P) Impulsive Behavior Scale. The secondary objective is to evaluate the safety of atomoxetine.

ELIGIBILITY:
Inclusion criteria

* Male and female subjects, 18-45 years of age at the time of consent meeting diagnostic criteria of Attention Deficit Hyperactivity Disorder (ADHD) per Diagnostic and Statistical Manual of Mental Disorders (DSM-5) at screening visit and currently undergoing diagnostic assessment and/or treatment for ADHD
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
* A diagnosis of the moderate symptoms of ADHD confirmed with combined score of 4 or higher in Clinical Global Impression-ADHD-Severity (CGI-ADHD-S) at Screening; Hyperactivity/Impulsivity subscale min 8 (at least moderate for impulsivity measure with ADHD checklist)
* Able and willing to discontinue the use of any psychotropic medications for treatment of ADHD symptoms, as well as of all relevant co-medication for comorbid conditions during the study
* Women of childbearing potential (WOCBP) [1] must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria and instructions on the duration of their use is provided in the patient information.

  1. A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Tubal ligation is NOT a method of permanent sterilisation.

Exclusion criteria

* Per DSM-5, had ever met diagnostic criteria for schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar disorder, delusional disorder or major depressive disorder (MDD) with psychotic features at the time of screening.
* Diagnosis of any mental disorder (according to DSM-5) that was primary focus of treatment within 6 months prior to Screening or at Baseline (as per clinical discretion of the investigator).

  --The following are not excluded: Substance Induced Mood Disorder, Major Depressive Disorder in remission, Generalized Anxiety Disorder in remission, Post-Traumatic Stress Disorder in remission, recreational/occasional substance use as long as willing to stop for duration of the study, Borderline Personality Disorder.
* Any psychiatric disorder, including the ones mentioned under #1, that in the opinion of the investigator would compromise participants' safety and/or validity of the data.
* Current or recent (in the 6 months prior to screening) suicidal ideation or behaviour of type 4 or 5 in the Columbia Suicidal Severity Rating Scale (C-SSRS).
* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR), temperature, or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator.
* Repeated measurement of systolic blood pressure outside the range of 90 to 145 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 45 to 90 mmHg, or pulse rate outside the range of 45 to 95 beats per minute (bpm).
* A marked baseline prolongation of QT/QTc interval ([QT/QTc = Time between start of the Q-wave and the end of the T-wave in an electrocardiogram / QT interval corrected for heart rate using the method of Fridericia (QTcF) or Bazett (QTcB)] such as QTc intervals that are repeatedly greater than 450 milliseconds (ms) in males or repeatedly greater than 470 ms in females) or any other relevant electrocardiogram (ECG) finding at screening.
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome).
* Further exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Rheinhessen-Fachklinik Alzey, Alzey
  - Universitätsklinikum Bonn AöR, Bonn
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Leipzig, Leipzig

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center, randomized, double-blind, placebo controlled parallel-group trial in participants with attention deficit hyperactivity disorder (ADHD). Eligible participants were randomized in a 1:1 ratio to receive either placebo or atomoxetine during a 2-week double-blind treatment period.
Pre-assignment Details: 63 male and female participants (32 atomoxetine, 31 placebo) were randomized and 62 participants were treated. Out of these, 58 completed the planned treatment and trial per protocol; 2 were erroneously randomized and discontinued (one treated and one not treated); 3 discontinued due to other reasons. All participants were free to withdraw at any time and were closely monitored.
Period: Overall Study
Arm/Group | Atomoxetine | Placebo (Matching Atomoxetine)
Started | 32 | 31
Number of Patients Treated | 31 | 31
Completed | 28 | 30
Not Completed | 4 | 1
Not completed — Not treated | 1 | 0
Not completed — Adverse Event | 2 | 1
Not completed — Exclusion criteria not met | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were treated with at least one dose of study drug (i.e. placebo or atomoxetine).
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo (Matching Atomoxetine) | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.4 (3.3) | 27.4 (4.4) | 26.4 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 16 | 14 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 22 | 48
  Unknown or Not Reported | 5 | 9 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 0 | 2
  White | 27 | 27 | 54
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Score of Barratt Impulsiveness Questionnaire v.11 (BIS-11) After Single Dose (at Day 1)
Description: The BIS-11 evaluates impulsiveness via 30 items scored on a 4-point scale (Rarely/Never = 1; Occasionally = 2; Often = 3; Almost Always/Always = 4). Total scores range from 30 (least impulsive) to 120 (most impulsive), calculated by summing item scores. Higher scores indicate greater impulsiveness.
  The data used in the analysis of covariance (ANCOVA) were estimated regardless of whether participants used rescue or other concomitant medications, or experienced nausea/vomiting. For participants who discontinued treatment early (receiving <90% of planned doses), their data were included in the analysis only up to the point of discontinuation.
  Reported summary data was based on an ANCOVA with the BIS-11 score at baseline as a covariate and the treatment arm as fixed factor.
Time Frame: Analysis based on the observation period: days 0 to 1, change from baseline calculated for Day 1.
Population: All randomized participants who received one dose of the study drug (placebo or atomoxetine) on Day 1 and had study data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Atomoxetine | Placebo (Matching Atomoxetine)
Number analyzed (Participants) | 30 | 31
Score on a scale | -0.8 [-2.3 to 0.8] | -0.4 [-1.9 to 1.1]
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo (Matching Atomoxetine); Change from baseline was analyzed with an ANCOVA model with the BIS-11 score at baseline as covariate and treatment as fixed factor; Test type: Other — No formal hypothesis was tested; ANCOVA; Least square mean difference = -0.4, 95% CI 2-sided [-2.6 to 1.7] — The treatment effect was estimated regardless of concomitant/rescue medication use or nausea/vomiting (treatment policy). Treatment discontinuation was handled with a while-on-treatment strategy

2. Primary Outcome: Change From Baseline in Total Score of Barratt Impulsiveness Questionnaire v.11 (BIS-11) at Steady State (at Day 14)
Description: as for outcome 1
Time Frame: Analysis based on the observation period: days 0 to 14, change from baseline calculated for Day 14.
Population: All randomized participants who received at least 90% (not more than one missed dose) of the planned doses of the study drug (placebo or atomoxetine) up to Day 14 and had study data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Atomoxetine | Placebo (Matching Atomoxetine)
Number analyzed (Participants) | 28 | 30
Score on a scale | -2.3 [-4.1 to -0.5] | -0.1 [-1.9 to 1.6]
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo (Matching Atomoxetine); [analysis description as in outcome 1, analysis 1]; Test type: Other — No formal hypothesis was tested; ANCOVA; Least square mean difference = -2.2, 95% CI 2-sided [-4.6 to 0.3] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Change From Baseline in Total Score of Short Urgency, Perseverance, Premeditation, and Sensation Seeking-Positive Urgency Impulsive Behavior Scale (S-UPPS-P) Impulsive Behavior Scale After Single Dose (at Day 1)
Description: The S-UPPS-P assesses impulsivity across five traits using 20 items scored on a 4-point scale (Agree Strongly = 1; Agree Some = 2; Disagree Some = 3; Disagree Strongly = 4). Total scores range from 20 (least impulsive) to 80 (most impulsive), calculated by summing item scores. Higher scores indicate greater impulsiveness.
  The data used in the analysis of covariance (ANCOVA) were estimated regardless of whether participants used rescue or other concomitant medications, or experienced nausea/vomiting. For participants who discontinued treatment early (receiving <90% of planned doses), their data were included in the analysis only up to the point of discontinuation.
  Reported summary data was based on an ANCOVA with the S-UPPS-P score at baseline as a covariate and the treatment arm as fixed factor.
Time Frame: Analysis based on the observation period: days 0 to 1, change from baseline calculated for Day 1.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Atomoxetine | Placebo (Matching Atomoxetine)
Number analyzed (Participants) | 30 | 31
Score on a scale | 0.0 [-1.6 to 1.6] | -0.1 [-1.7 to 1.4]
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo (Matching Atomoxetine); Change from baseline was analyzed with an ANCOVA model with the S-UPPS-P score at baseline as covariate and treatment as fixed factor; Test type: Other — No formal hypothesis was tested; Least square mean = 0.2, 95% CI 2-sided [-2.1 to 2.4] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Change From Baseline in Total Score of Short Urgency, Perseverance, Premeditation, and Sensation Seeking-Positive Urgency Impulsive Behavior Scale (S-UPPS-P) Impulsive Behavior Scale at Steady State (at Day 14)
Description: as for outcome 3
Time Frame: Analysis based on the observation period: days 0 to 14, change from baseline calculated for Day 14.
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Atomoxetine | Placebo (Matching Atomoxetine)
Number analyzed (Participants) | 28 | 30
Score on a scale | -0.2 [-1.7 to 1.4] | -1.0 [-2.5 to 0.5]
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo (Matching Atomoxetine); [analysis description as in outcome 3, analysis 1]; Test type: Other — No formal hypothesis was tested; ANCOVA; Least square mean difference = 0.9, 95% CI 2-sided [-1.3 to 3.1] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Patients With Treatment Emergent Adverse Events and Serious Adverse Events
Description: Treatment emergent adverse events are adverse events that occurred after treatment administration up to 4 days after the last dose of study drug.
Time Frame: From first drug administration on Day 1 until Day 16 + 4 days (REP), up to 20 days.
Population: All participants who were treated with at least one dose of study drug (i.e. placebo or atomoxetine).
Measure: Number; unit: Percentage (%) of participants
Arm/Group | Atomoxetine | Placebo (Matching Atomoxetine)
Number analyzed (Participants) | 31 | 31
Percentage (%) of participants
  Treatment-emergent adverse events | 90.3 | 80.6
  Treatment-emergent serious adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events: From first drug administration on Day 1 until Day 16 + 4 days (REP), up to 20 days. All-cause mortality: From first drug administration on Day 1 until Day 28, up to 28 days.
Description: Treated Set (TS): All subjects who were treated with at least one dose of study drug (i.e. placebo or atomoxetine)
Arm/Group | Atomoxetine | Placebo (Matching Atomoxetine)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 28/31 | 23/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atomoxetine (N=31) | Placebo (Matching Atomoxetine) (N=31)
Palpitations (Cardiac disorders) | 5 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 14 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Fatigue (General disorders) | 8 | 5
Feeling cold (General disorders) | 2 | 0
Feeling hot (General disorders) | 3 | 0
Nasopharyngitis (Infections and infestations) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 10 | 0
Disturbance in attention (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 9 | 1
Headache (Nervous system disorders) | 13 | 9
Paraesthesia (Nervous system disorders) | 3 | 0
Apathy (Psychiatric disorders) | 4 | 1
Initial insomnia (Psychiatric disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 2 | 2
Irritability (Psychiatric disorders) | 2 | 1
Sleep disorder (Psychiatric disorders) | 3 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT05278104/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT05278104/SAP_001.pdf